CLINICAL TRIAL: NCT00732485
Title: The Role of Mitochondrial Oxidation on Insulin Resistance in Burn Patients Treated With Fenofibrate
Brief Title: Mitochondrial Oxidation and Insulin Resistance in Burn Patients Treated With Fenofibrate
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Principal Investigator Changed
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Shriners Hospitals for Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-389; SHC 08-GAL-006
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Burn
Keywords: Burn injury; Fenofibrate; Insulin resistance; Mitochondrial function; Fat oxidation; PPAR; Protein; Glucose; Wound
MeSH Terms: conditions — Burns; Insulin Resistance; Wounds and Injuries | interventions — Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fenofibrate (Active Comparator)
  Interventions: Drug: fenofibrate
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: fenofibrate — Fenofibrate, PO, 5 mg/kg/day from admission to 6 months post burn
  Arms: Fenofibrate
Drug: placebo — Placebo, sugar pill, from admission to 6 months post burn
  Arms: Placebo

SUMMARY:
Major burn injury causes significant insulin resistance on glucose and protein metabolism that persists for up to 6 months after the acute injury

This project proposes to answer the following questions:

1. Will fenofibrate given to burn patients with insulin resistance restore their insulin sensitivity?
2. What is the relationship between mitochondrial dysfunction in muscle tissue as the causative mechanism of burn related insulin resistance?
3. To what extent will the restored insulin sensitivity affect glucose and protein metabolism in muscle, regenerating wounds and the liver, i.e. ameliorate burn related hyperglycemia and protein catabolism?

DETAILED DESCRIPTION:
The following specific hypotheses will be investigated:

1. Following severe burn injury in human patients the mitochondrial fat oxidation capacity is decreased in muscle. This is associated with a corresponding progression in the severity of the resistance to the action of insulin on glucose disposal and protein synthesis and breakdown in muscle, regenerating wound and liver.
2. Fatty acids, or their active intracellular products (e.g., DAG, acyl-CoenzymeA (Co-A), or acylcarnitine), are the direct inhibitors of insulin action, rather than tissue triglycerides (TG) itself. In other words, impaired mitochondrial fatty acid oxidation is the mechanism that causes altered lipid metabolism that ultimately contributes to insulin resistance.
3. Accumulation of active fatty acid products, such as DAG, acyl-CoA, or acylcarnitine esters in muscle cells is due to the rate of uptake of plasma free fatty acid (FFA) exceeding the rate of oxidation within muscle due principally to a reduced capacity of mitochondria to oxidize fatty acids.
4. Decreased insulin sensitivity in muscle is related to impaired insulin signaling. This will be reflected by increased activity of protein kinase C (PKC). Because PKC is thought to exert its regulatory effect primarily on either tyrosine kinase activity on the insulin receptor or downstream kinase insulin receptor substrate (IRS) phosphorylation, these elements of the insulin signaling cascade will be decreased. In turn, elements of insulin signaling related to the response of muscle glucose (PI3 kinase) and protein (P70S6k) metabolism will be reduced. We propose that increased tissue PKC activity will be associated with increased tissue concentration of DAG, acyl-CoA, or acylcarnitine.
5. Treatment of patients with the peroxisome proliferator-activated receptor (PPAR) alpha agonist fenofibrate will improve mitochondrial capacity to oxidize fatty acids.
6. Insulin sensitivity in muscle, skin and liver in terms of both glucose and protein metabolism will be improved by fenofibrate treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 7 years old with burns covering 40% or more of body surface who are admitted to the Shriners Hospital for Children, Galveston, Texas

Exclusion Criteria:

* Abnormal liver and kidney function,
* Pregnancy,
* Diabetes mellitus,

Ages: 7 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity on glucose and protein metabolism | From admission to burn unit to 6 months post burn

SECONDARY OUTCOMES:
Systemic glucose homeostasis | Admission to 6 months post burn
Muscle protein balance | Admission to 6 months post burn
Wound protein balance | Admission to 6 months post burn

CONTACTS AND LOCATIONS:
Overall Officials: David Herndon, MD, Principal Investigator — University of Texas Medical Branch, Galveston

REFERENCES:
- [Result] Cree MG, Zwetsloot JJ, Herndon DN, Qian T, Morio B, Fram R, Sanford AP, Aarsland A, Wolfe RR. Insulin sensitivity and mitochondrial function are improved in children with burn injury during a randomized controlled trial of fenofibrate. Ann Surg. 2007 Feb;245(2):214-21. doi: 10.1097/01.sla.0000250409.51289.ca. PMID 17245174